CLINICAL TRIAL: NCT06446180
Title: Streptococcus Salivarius K12@Lip@GSH preventsOral Mucositis in Patients Undergoingintensity Modulated Radiotherapy for Malignant Head and Neck Tumors(Including Nasopharyngeal Carcinoma) : A Single, Single Arm Prospective Trial
Brief Title: Streptococcus Salivarius K12@Lip@GSH Alleviates Oral Mucositis in Patients Undergoing Radiotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Responsible Party: Principal Investigator, Zhihui Li, PhD,Professor, The General Hospital of Western Theater Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-002
Record Dates: First submitted 2024-05-09; First posted 2024-06-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): SsK12@Lip@GSH
  Interventions: Drug: SsK12@Lip@GSH

INTERVENTIONS:
Drug: SsK12@Lip@GSH — SsK12@Lip@GSH powder contained 1×10^9 CFU viable cells of SsK12@Lip@GSH as the active ingredient.

SUMMARY:
Radiation-induced oral mucositis (RIOM) is the most common oral complication of cancer patients receiving radiotherapy and/or chemotherapy, leading to poor quality of life. the investigators previous studies that have reported the use of single SSK12 probiotics in RIOM. However, SSK12 probiotics alone may lack stability, free radical scavenging activity and oral local targeting.Here, the investigators designed a new oral probiotic K12@Lip@GSH that SSK12 is encapsulated in liposomes(Lip) to enhance its stability and free radical scavenging ability, and glutathione (GSH) transporter-mediated oral targeting agent based on the over-expression of GSH transporters at the RIOM. The investigators have complete evaluated the treatment outcome of SSK12@Lip@GSH on RIOM mice.

The investigators designed a single-center, single-arm prospective clinical study to evaluate the safety and efficacy of SsK12@Lip@GSH in the treatment of radioactive oral mucositis in patients with head and neck malignancies

DETAILED DESCRIPTION:
Radiotherapy (RT) is an important method of treatment for malignant tumors of the head and neck and can be used alone or in combination with chemotherapy as a radical or adjuvant therapy. Despite improvements in RT equipment and techniques, various acute oral complications persist, including oral mucositis (OM), dry mouth, taste dysfunction, and oral infections. OM is one of the most common acute radiation-related toxicities, and approximately 50%-70% of patients experience severe OM (SOM) defined by the WHO scale as grade 3 to 4. The painful inflammation and ulceration associated with OM not only profoundly affect patients' ability to eat, swallow, and speak, but also decrease their tolerance to anti-cancer treatment, thereby, impairing their quality of life (QoL) significantly and causing interruptions in their cancer treatment. Although some clinical strategies for radiation-induced OM have been recommended by the Multinational Association of Supportive Care in Cancer and the International Society of Oral Oncology (MASCC/ISOO) , their efficacy and safety still need further clinical validation. Recent evidence suggests the involvement of oral microbiota in radiationinduced OM, and modulation of oral microbiota is promising for the management of OM. Streptococcus salivarius K12 is a commercially available oral probiotic with strong oral colonization ability, bacteriocin-like inhibitory substance (BLIS)-producing capability, and immunomodulatory properties, and has been used to treat oral candidiasis, pharyngitis, tonsillitishalitosis, and otitis media. More importantly, data from our recent animal study demonstrated that topical use of S. salivarius K12 ameliorates radiationinduced OM in mice by modulating the oral microbiota, mainly by suppressing oral anaerobes.

the investigatorsprevious studies that have reported the use of single SSK12 probiotics in RIOM. In 2024, the applicant team published a randomized controlled trial as the first author in the top journal in the field of oncology, Journal o f Clinical Oncology, which found that Streptococcus salivarius K12 (SSK12) can effectively alleviate RIOM in radiotherapy patients with malignant head and neck tumors.

However, SSK12 probiotics alone may lack stability, free radical scavenging activity and oral local targeting.Here, the investigators designed a new oral probiotic K12@Lip@GSH that SSK12 is encapsulated in liposomes(Lip) to enhance its stability and free radical scavenging ability, and glutathione (GSH) transporter-mediated oral targeting agent based on the over-expression of GSH transporters at the RIOM. the investigators evaluated the treatment outcome of SSK12@Lip@GSH on RIOM mice .

In vitro studies showed that SSK12@Lip@GSH treatment was beneficial for the healing of RIOM mice, as reflected by reduced ulcer size, increased basal layer epithelial cellularity and mucosal thickness, and elevated epithelial proliferation and attenuated apoptosis. Genomic results showed that the SSK12@Lip@GSH could improve relevant mRNA pathways to promote RIOM healing. In addition, SSK12@Lip@GSH treatment reconstituted the oral microbiota and decreased the abundance of oral anaerobes of RIOM mice.Therefore, the SSK12@Lip@GSH holds promise as a potential approach for preventing and treating radiation-induced oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
* 2. Aged 18-80 years;
* 3. Eastern Cooperative Oncology Group performance status of ≤2;
* 4. Planning to receive definitive RT or postoperative adjuvant RT;
* 5. Normal liver, kidney and bone marrow function;
* 6. Sign informed consent.

Exclusion Criteria:

* 1.Known hypersensitivity or more severe allergies to Lactobacillus Reuteri components;
* 2.Those with poor compliance;
* 3.Pregnancy or breastfeeding;
* 4.History of head and neck radiotherapy;
* 5.Taking antifungal or viral medications one week prior to the start of radiation therapy.
* 6.Other patients (with any other serious other medical condition) who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
The incidence of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale.The WHO Oral Toxicity Scale categorizes oral mucositis into grades 0-4, with the higher the grade the more severe the patient's oral mucositis. Grade 0 means that the oral mucosa is normal and the patient has no symptoms or signs; grade 1 means that the mucosa is erythematous with or without pain and does not interfere with eating; grade 2 means that the mucosa is erythematous and ulcerated, but still able to eat solid food; grade 3 means that the mucosa is severely ulcerated with extensive erythema and unable to eat solid food; and grade 4 means that the ulcers of the mucosa are fused together into a sheet, and their severity is so severe that it is not possible to eat.

SECONDARY OUTCOMES:
The time to onset of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Time from the first day of radiotherapy to the first determination of SOM. Patients without observed SOM were assigned onset days of 6 or 6.5 weeks
The duration of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM. Patients without observed SOM were assigned a duration of 0 days
Mouth and throat soreness (MTS) scores | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms
Xerostomia summated xerostomia inventory (SXI) | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Xerostomia is subjectively assessed on the Summated Xerostomia Inventory (SXI). The SXI is categorized according to score as 0 no dry mouth (5), 1 mild dry mouth (6-8), 2 moderate dry mouth (9-12), and 3 severe (13-15).
Functional assessment of cancer therapy-head and neck (FACT- H&N) quality of life questionnaire | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  FACT- H&N quality of life questionnaire 4.0 is a scale used to assess quality of life in
Adverse events | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version
Oral activities scores | From the start of radiotherapy to 4 weeks after completion of radiotherapy
  Patients report the degree to the impact of MTS on oral activities (including swallowing, drinking, eating, talking, sleeping) (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: zhihui li, Principal Investigator — The General Hospital of Western Theater Command
Locations (1):
- Department of Oncology，The General Hospital of Western Theater Command, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No